CLINICAL TRIAL: NCT02179333
Title: Preliminary Study of the Scale To Assess Ataxia and Neurologic Dysfunction (STAND)
Acronym: STAND
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Theresa Zesiewicz, MD, Professor of Neurology, University of South Florida
Other Study IDs: STAND2012
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Spinocerebellar Ataxia - All Sub-types; Friedreich's Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with Ataxia: Patients with a diagnosis of ataxia (Friedreich's ataxia or Spinocerebellar ataxia type 1-30) aged 18-80 years old will be recruited for the study.
  Interventions: Other: Ataxia rating scale

INTERVENTIONS:
Other: Ataxia rating scale — Administer new rating scale for ataxia. This will be administered by two different raters on two separate occassions, 4 to 6 weeks apart.

SUMMARY:
The objectives of this study are:

* To validate the inter-rater and intra-rater reliability of a new scale for the assessment of ataxia and neurologic dysfunction (STAND)
* To assess common constructs and correlation between STAND subscale items.

DETAILED DESCRIPTION:
There are few validated, comprehensive rating scales for the assessment of ataxia severity. The development of a Scale To assess Ataxia and Neurologic Dysfunction (STAND) would examine and measure as many facets of ataxia as possible. Scale items to be measured include parkinsonism, timed gait analysis, dystonia, neuropathy and peripheral nerve weakness, as well as other areas of clinical manifestation for ataxia. This brief but thorough scale should yield a thorough measurement of ataxia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ataxia.
* Male or female between 18 and 80 years of age.
* Subject has voluntarily signed an IRB approved informed consent form to participate in the study after all relevant aspects of the study have been explained and discussed with the subject.

Exclusion Criteria:

* Any illness that in the investigator's opinion preclude participation in this study.
* Subjects with a cardiac pacemaker
* Legal incapacity or limited legal capacity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community members, support group members or clinic patients with ataxia.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Inter- and intra-rater agreement | 4 to 6 weeks
  Assess agreement between raters (inter-rater agreement) and within raters (intra-rater agreement) through the evaluation of STAND total score, subtotals and individual variables using intraclass correlation coefficients (ICCs).

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States